CLINICAL TRIAL: NCT07135310
Title: STROKE 120 ACTION: a National Cluster Randomized Controlled Trial
Brief Title: STROKE 120 ACTION Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Minhang Central Hospital (Other)
Responsible Party: Principal Investigator, Jing Zhao, Chief of the Department of Neurology, Shanghai Minhang Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-055-01K
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Pre-hospital delay; Cluster-randomized trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Usual health policy plus STROKE 120 multifaceted intervention campaign
  Interventions: Behavioral: STROKE 120 multifaceted intervention campaign
- Control group (No Intervention): Usual health policy alone

INTERVENTIONS:
Behavioral: STROKE 120 multifaceted intervention campaign — Based on the existing usual health policy, the intervention group will implement a STROKE 120 multifaceted intervention campaign in the intervention community units for a continuous period of 12 months (3-month intensive period and 9-month maintenance period).
  The detailed implementation plan for the STROKE 120 multifaceted intervention campaign in the intervention group is as follows:
  1. Training medical workers in stroke center;
  2. Training emergency center staff and primary care physicians;
  3. Conducting public education;
  Arms: Intervention group

SUMMARY:
Stroke is the main cause of death and disability in China, but it is preventable and treatable. For the most common type, acute ischemic stroke (AIS), initiating reperfusion therapy with intravenous thrombolysis (IVT) with or without mechanical thrombectomy (MT) within several hours of the onset of symptoms can significantly improve the chances of surviving free of major disability, and earlier the intervention is given the better the outcome. Thus, whether patients can achieve timely arrived at hospital, ideally within the critical 4.5-hour golden window, is pivotal to achieving high rates of recanalization and optimal functional outcome. To this end, it is important to note that the overall pre-hospital delay for patients with AIS is currently 24 hours in China.

We plan to conduct STROKE 120 ACTION, a national cluster randomized controlled trial, to determine whether implementing a STROKE 120 multifaceted intervention campaign can reduce pre-hospital delay in AIS, increase the 4.5-hour hospital arrival rate, and improve survival, disability, and healthcare costs. The STROKE 120 ACTION trial will recruit 16 community units across 8 regions in China, with each region enrolling 2 community units with a residential population of at least 110,000 and comparable demographic characteristics. To avoid cross-contamination, the participating community clusters will maintain a physical distance of more than 20 kilometers. Within each region, the 2 community units will be randomly assigned at a 1:1 ratio to receive the intervention (12-month usual health policy plus STROKE 120 multifaceted intervention campaign; 3-month intensive period and 9-month maintenance period) or control (12-month usual health policy alone). The study outcomes and related data on incident AIS cases within each participating community unit will be collected after the implementation of STROKE 120 multifaceted intervention campaign (from month 1 to month 12 of multifaceted intervention campaign). The primary outcome is proportion of hospital arrival within 4.5 hours after symptom onset within participating community units. Secondary outcomes include time from onset to hospital admission, time from onset to action, use of 120 emergency ambulances, IVT, MT, total hospitalization costs, out-of-pocket costs, composite outcome of death or major disability (modified Rankin scale score [mRS] ≥3) at 3 months, ordinal 7-level mRS score at 3 months, all-cause mortality within 3 months. The sample size was calculated according to the following estimates: (1) a significance level of 0.05 for a 2-sided test; (2) statistical power of 85%; (3) 4.5-hour hospital arrival rate of 10% for AIS patients in control group; (4) 4.5-hour hospital arrival rate of 20% among AIS patients in intervention group; (5) intra-class correlation coefficient of 0.03; and (6) a 10% loss to follow-up. The estimated sample size is 3,312 incident AIS patients from 16 community units with an average cluster size of 207 patients per community unit. The annual incidence of AIS is 195 per 100,000 people, and the sample size of participants in each community unit will be 106,000. Thus, the total sample size of the present study will be 1,696,000 participants from 16 community units.

The STROKE 120 ACTION trial will address the critical issue of long pre-hospital delay in AIS in China, and provide profound implications for global stroke prevention and control strategies.

ELIGIBILITY:
This trial will evaluate whether the STROKE 120 multifaceted intervention campaign can reduce the pre-hospital delay in AIS and increase the 4.5-hour arrival rate in 16 community units across 8 regions in China. We will select 2 community units from each region as the study sites and randomly divide the 2 community units within each region into the intervention group and the control group. The selection criteria for community units are listed as follows:

1. The 2 participating community units in each region should each have a permanent population over 110,000 (people aged 60 years and above accounting for at least 15%), have similar demographic characteristics (e.g., age, gender, and education level), and have comparable local health policies (e.g., medical insurance policies, emergency system framework, stroke emergency map release, and stroke center quality control), economic levels, and public ability to recognize AIS.
2. The participating hospitals in each community unit serve >90% of AIS patients within the community unit, have a well-established stroke center, and have comparable standardized treatment capabilities for AIS (including 4.5-hour hospital arrival rate of AIS, rate of using 120 emergency ambulances after AIS, and rate of IVT after AIS).
3. The participating communities are capable of implementing STROKE 120 multifaceted intervention campaign within its community unit.
4. To avoid cross-contamination, the physical distance between any two community units exceeds 20 kilometers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1696000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Arriving hospital within 4.5 hours after symptom onset among incident acute ischemic stroke cases within participating community units | From month 1 to month 12 of multifaceted intervention campaign
  Proportion of arriving hospital within 4.5 hours after symptom onset among incident acute ischemic stroke cases within participating community units

SECONDARY OUTCOMES:
Time from onset to hospital admission after acute ischemic stroke | From month 1 to month 12 of multifaceted intervention campaign
Time from onset to action after acute ischemic stroke | From month 1 to month 12 of multifaceted intervention campaign
Use of 120 emergency ambulances after acute ischemic stroke | From month 1 to month 12 of multifaceted intervention campaign
  Proportion of using 120 emergency ambulances after acute ischemic stroke
Intravenous thrombolysis after acute ischemic stroke | From month 1 to month 12 of multifaceted intervention campaign
  Proportion of intravenous thrombolysis after acute ischemic stroke
Mechanical thrombectomy after acute ischemic stroke | From month 1 to month 12 of multifaceted intervention campaign
  Proportion of mechanical thrombectomy after acute ischemic stroke
Total hospitalization costs | At Hospital Discharge after ischemic stroke onset (ischemic stroke patients occurring from month 1 to month 12 of multifaceted intervention campaign)
Out-of-pocket hospitalization costs | At Hospital Discharge after ischemic stroke onset (ischemic stroke patients occurring from month 1 to month 12 of multifaceted intervention campaign)
Composite outcome of death or major disability at 3 months after acute ischemic stroke | Three months after ischemic stroke (ischemic stroke patients occurring from month 1 to month 12 of multifaceted intervention campaign)
  The composite outcome of death or major disability was defined as a score of 3 to 6 on the modified Rankin Scale at 3 months after ischemic stroke. Scores on the modified Rankin Scale range from 0 to 6, with a score of 0 indicating no symptoms; a score of 5 indicating severe disability (ie, bedridden, incontinent, or requiring constant nursing care and attention); and a score of 6 indicating death.
Ordinal 7-level modified Rankin Scale score at 3 months after acute ischemic stroke | Three months after ischemic stroke (ischemic stroke patients occurring from month 1 to month 12 of multifaceted intervention campaign)
  Scores on the modified Rankin Scale range from 0 to 6, with a score of 0 indicating no symptoms; a score of 5 indicating severe disability (ie, bedridden, incontinent, or requiring constant nursing care and attention); and a score of 6 indicating death.
All-cause mortality within 3 months after acute ischemic stroke | Three months after ischemic stroke (ischemic stroke patients occurring from month 1 to month 12 of multifaceted intervention campaign)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Minhang Central Hospital, Shanghai, China